CLINICAL TRIAL: NCT04383132
Title: Does Using Abdominal Binder Really Benefit During Colonoscopy ?: A Prospective, Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Effectiveness of Abdominal Binder Use During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Beslen Goksoy, Principal Investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Beslen-korse
Record Dates: First submitted 2020-05-04; First posted 2020-05-12 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Performance and Tolerance of Colonoscopy
Keywords: abdominal binder; colonoscopy; loop

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Binder Intervention Group (Experimental): Patients randomized to Abdominal Binder Intervention Group will have the abdominal binder secured firmly between Spina iliaca anterior superior and subcostal area to the abdomen just prior the colonoscopy.
  Interventions: Device: Abdominal Binder
- Sham Group (Sham Comparator): Sham Group will have the abdominal binder secured firmly between Spina iliaca anterior superior and subcostal area to the abdomen just prior the colonoscopy but it will be loosened just prior the procedure
  Interventions: Device: Abdominal Binder

INTERVENTIONS:
Device: Abdominal Binder — abdominal binder is a kind of elastic abdominal compression device

SUMMARY:
Colonoscopy is considered the primary screening test for colorectal cancer screening worldwide. For technical difficulties previously experienced during colonoscopy, especially loop of the colonoscopy device in the colon, many solution methods have been developed and applied (manual pressure and position change, etc.). Although these methods are partially successful, there is no consensus on the optimum solution method. Few studies in the literature have investigated the use of corset during colonoscopy and conflicting results have been reported. In this study, elastic abdominal corset or false corset will be used during colonoscopy. Indeed, the investigators aim to determine whether this method is effective and safe with their own results and contribute to the literature. The primary outcome of this study will be the cecal intubation time. Secondary outcomes include manual pressure and position change during the procedure, length of cecal intubation (length of colonoscope required to reach the cecum from the anus), colonoscopy completion rate, additional anesthesia and / or analgesic requirement, patient pain and comfort level and colonoscopic findings.Efficacy will be assessed on the basis of pairwise comparisons between groups with respect to primary and secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

Between the ages of 18 - 90 Participants must have completed the full prescribed colonoscopy purgative preparation prior to their procedure, and describe adequate cleansing.

Participants with ASA I-III (American Society of Anesthesiologists Class III)

Exclusion Criteria:

Previous colon resection History of intra-abdominal malignancy Known anesthetic or analgesic drugs allergy Multiple planned procedures (e.g.bidirectional endoscopy) Pregnancy Active inflammatory bowel disease A history of intraabdominal malignancy History of cirrhosis or ascites Known ventral hernia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beslen Göksoy, M.D., Principal Investigator — Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Locations (1):
- Martyr Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Starting 6 months after publication

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Started | 173 | 173
Completed | 173 | 173
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abdominal Binder Intervention Group | Sham Group | Total
Number analyzed (Participants) | 173 | 173 | 346
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.53 (12.3) | 52.57 (12.41) | 51.55 (12.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 108 | 205
  Male | 76 | 65 | 141
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 173 | 173 | 346
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.79 (5.02) | 29.62 (5.54) | 29.2 (5.3)
waist circumference (WC) [Mean (Standard Deviation); unit: cm] | 102.33 (10.67) | 103.26 (11.84) | 102.8 (11.27)

OUTCOME MEASURES:

1. Primary Outcome: Mean Cecal Intubation Time
Description: Cecal intubation time will be defined as the time from insertion of the colonoscope into the rectum to identification of the base of the cecum
Time Frame: During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified,an average of 1-30 minutes
Population: 9 patients were excluded from analysis CIT and CIL because the incompleted procedure (intervention group n 4, sham group n 5). Because the procedure must be completed for CIT and CIL analysis.
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 169 | 168
sec | 240 (110) | 250 (115)
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; In sample size calculation, CIT and SD were used. It was found that 326 patients (163 per group) were required to detect a 60-second difference in CIT (SD 192 secs), with 80% power and two-sided alpha 0.05. The frequency of the auxiliary maneuvers was calculated that 324 patients were required for a 20% reduction in the auxiliary maneuvers. In case of becoming lost to follow up and withdrawal, the number of patients was expanded by 5%, and a total of 346 patients, were included in the study; Test type: Other; p = 0.388, t-test, 2 sided — Independent t-test was used to compare mean CIT between two groups. The statistical significance level was accepted as p<0.05

2. Secondary Outcome: Number of Participants Who Required Ancillary Maneuvers
Description: Binary data indicating individually whether abdominal pressure or patient position change was used during the insertion phase of the procedure will be recorded.
Time Frame: During colonoscopy, from insertion of scope into rectum to point in time when base of cecum is identified, an average of 1-30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 173 | 173
Participants | 65 | 85
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.069, Chi-squared — For the comparison of ancillary maneuvers Pearson chi-square test, Fisher's exact test, and Fisher-Freeman-Halton exact test were used

3. Secondary Outcome: Length of Cecal Intubation
Description: The length of the colonoscope required to reach the cecum from the anus will be measured
Time Frame: From inserting the scope into the rectum during the colonoscopy, until the cecum base is determined, an average of 1-30 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 169 | 168
cm | 89 (18) | 88.5 (15)
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.487, t-test, 2 sided — Independent t-test was used to compare mean CIL between two groups

4. Secondary Outcome: Number of Participants Who Completed the Procedure
Description: Dichotomous outcome indicating if the procedure was incomplete or complete.
Time Frame: During colonoscopy, from time point of insertion of scope into rectum to point in time when scope is removed from rectum,an average of 2-60 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 173 | 173
Participants | 169 | 168
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.822, Chi-squared

5. Secondary Outcome: Number of Participants Who Required Additional Anesthetic and / or Analgesic Drug
Description: Whether the patient needs an additional dose of anesthetic and / or analgesic drug to complete the colonoscopy
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 173 | 173
Participants | 43 | 64
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.016, Chi-squared

6. Secondary Outcome: Patient Pain and Comfort Level at Discharge
Description: Study assistant will interview patient just prior to discharge and obtain responses for pain according to 10-point visual analog scales ( scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" =1 (min) and "worst pain"=10 (max)) and global satisfaction according to a 5-point scale ( scores are recorded by making a handwritten mark on a 5-cm line that represents a continuum between "very unsatisfied" =1 (min) and "very satisfied"=5 (max) )
Time Frame: At single time point occurring after the colonoscopy, just prior to the patient being discharged from facility,an average of 60 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 173 | 173
score on a scale
  VAS score | 1.9 (1.6) | 3.3 (1.8)
  patient satisfaction score | 1.7 (0.9) | 1.7 (0.9)
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.001, t-test, 2 sided

7. Secondary Outcome: Number of Participants According to Colonoscopy Findings
Description: Findings such as polyp, cancer, diverticulum detected during colonoscopy will be recorded.
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Abdominal Binder Intervention Group | Sham Group
Number analyzed (Participants) | 173 | 173
Participants
  Polyps | 72 | 70
  Diverticulosis | 60 | 59
  No mucosal pathology | 38 | 42
  IBD or colitis | 0 | 2
  colon cancer | 3 | 0
Statistical Analysis 1: Comparison: Abdominal Binder Intervention Group vs Sham Group; Test type: Other; p = 0.184, Fisher Exact

ADVERSE EVENTS:
Time Frame: Time from the start of the colonoscopy until the patient's discharge, approximately 1-2 hours
Arm/Group | Abdominal Binder Intervention Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/173
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/173
Other Adverse Events (participants affected / at risk) | 0/173 | 0/173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04383132/Prot_SAP_ICF_000.pdf